CLINICAL TRIAL: NCT01871376
Title: Intravitreal Aflibercept Injection for Polypoidal Choroidal Vasculopathy With Hemorrhage or Exudation
Acronym: EPIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gregg T. Kokame, MD (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Gregg T. Kokame, MD, Primary Investigator, Hawaii Pacific Health
Organization: Hawaii Pacific Health (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIC
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: PCV
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Previously Treated (Active Comparator): Patients that have previously received treatment for polypoidal choroidal vasculopathy.
  Intervention: Monthly 2.0mg intravitreal aflibercept injection, followed by Q8W dosing with 2.0mg intravitreal aflibercept injection or as often as monthly if needed for 1 year for previously treated arm.
  Interventions: Drug: Intravitreal aflibercept injection 2.0mg
- Treatment-Naive (Active Comparator): Patients that have not received treatment for polypoidal choroidal vasculopathy.
  Intervention: Monthly 2.0mg intravitreal aflibercept injection, followed by Q8W dosing with 2.0mg intravitreal aflibercept injection or as often as monthly if needed for 1 year for treatment-naive arm.
  Interventions: Drug: Intravitreal aflibercept injection 2.0mg

INTERVENTIONS:
Drug: Intravitreal aflibercept injection 2.0mg — Monthly 2.0mg intravitreal aflibercept injection, followed by Q8W dosing with 2.0mg intravitreal aflibercept injection or as often as monthly if needed for 1 year for both treatment naive and prior treatment arms.
  Other Names: Eylea

SUMMARY:
To evaluate the efficacy and safety of intravitreal aflibercept injection in the treatment of PCV

DETAILED DESCRIPTION:
This is an open-label, randomized, one-year, multiple-dose study of 2mg aflibercept in patients with PCV.

The study consists of the baseline visit on day 0 and a mandatory clinic visit every 30 days to assess efficacy and safety. All patients will receive three monthly injections of 2mg intravitreal aflibercept injection followed by treatment every 60 days through 720 days (24 months). Patients can be treated every 30 days if needed.

The fellow eye may be treated with intravitreal aflibercept injection per the investigator's discretion at any point during the study if evidence of disease activity are met: exudation or hemorrhage secondary to polypoidal choroidal vasculopathy or exudative AMD. The fellow eye will not be considered the study eye. If treatment with aflibercept is to be given in the fellow eye, the injections are to be administered according to the Food and Drug Administration (FDA) approved label for EYLEA®.

ELIGIBILITY:
Inclusion Criteria:

* Age > 25 years of age.
* In the opinion of the principal investigator, the study eye has PCV with active exudation and/or bleeding that may benefit from treatment with study medication.
* Diagnosis of PCV via ICG Angiography with evidence of active leakage, active bleeding or recent decreased in vision.
* Baseline visual acuity better than or equal to 20/200 using ETDRS
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent

Exclusion Criteria:

* Any history of previous vitrectomy
* Previous cataract surgery within the preceding 2 months of Day 0
* Active infections conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Presence of any condition that would jeopardize the patient's participation in this study
* Participation in an investigational trial within 30 days of randomization that involved treatment with any drug that has not received regulatory approval at the time of study entry
* For the Treatment-Naïve cohort: no prior anti-VEGF (Macugen, Avastin, Lucentis, Eylea) in the study eye
* For the Previous-Treated cohort: no prior anti-VEGF (Macugen, Avastin, Lucentis) in the study eye within 30 days or enrollment in this study
* For the Previous-Treated cohort: no prior Eylea in the study eye
* Known allergy to any component of the study drug
* Blood pressure >180/119 (systolic above 180 or diastolic above 110). If blood pressure is brought below 180/110 by anti-hypertensive treatment, the patient can be eligible.
* Major surgery within 28 days prior to randomization or major surgery planned within the next 12 months. Major surgery is defined as a surgical procedure that is more extensive than needle biopsy/aspiration placement of a central venous access device, removal/biopsy of a skin lesion, or placement of a peripheral venous catheter
* Myocardial infarction, other cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 6 months prior to randomization
* Systemic anti-VEGF or pro-VEGF treatment within 3 months prior to randomization
* Pregnant or breast-feeding women
* Simultaneous participation in another medical investigational trial
* Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly)

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
efficacy of intravitreal aflibercept injection of 2.0mg aflibercept | 2 Years
  This study will evaluate the efficacy of intravitreal aflibercept injection of 2.0mg aflibercept administered Q8W following an initial loading dose of 3 monthly injections in patients with polypoidal choroidal vasculopathy with active exudation or bleeding as measured by:
  • Mean change in BCVA between Day 0 (Baseline) and Day 720 (M24)

SECONDARY OUTCOMES:
Proportion of Patients with Stable, Improved, Significant Improved, Decreased, Significant Decreased Vision | 6 Months, 12 Months, 18 Months, 24 Months
  To evaluate the proportion of patients at Day 180 (M6), Day 360 (M12), Day 540 (M18) and Day 720 (M24) with "Stable" vision <5 letters gained or lost, "Improved" vision >5 letters gained, "Significant Improved" vision ≥15 letters gained, "Decreased" vision >5 letters lost, "Significant Decreased" vision ≥15 letters lost
Proportion of Patients with decrease in Subretinal Hemorrhage and/or Exudates | Month 6, Month 12, Month 18, Month 24
  To evaluate the proportion of patients at Day 180 (M6), Day 360 (M12), Day 540 (M18), Day 720 (M24) in decreasing subretinal hemorrhage and/or subretinal exudates via fundus photos and fundus exams
Proportion of patients with decreased / complete resolution of Polypoidal Polyp. | Month 3, Month 6, Month 12, Month 18, Month 24
  To evaluate the proportion of subjects with a decrease and/or complete resolution of polypoidal polyps from PCV at Day 90 (M3), Day 180 (M6), Day 360 (M12), Day 540 (M18) and Day 720 (M24) as assessed by fluorescein and indocyanine green angiography
Proportion of subject with a decrease or complete resolution of branching vascular network from PCV | Month 3, Month 6, Month 12, Month 18, Month 24
  To identify the proportion of subjects with a decrease and/or complete resolution of branching vascular network (BVN) from PCV at Day 90 (M3), Day 180 (M6), Day 360 (M12), Day 540 (M18) and 720 (M24) months as assessed by fluorescein and indocyanine green angiography
Determine mean change in Central Foveal Thickness and/or peripapillary edema as measured by SD-OCT | Baseline, Month 6, Month 12, Month 18, Month 24
  To determine mean change in central foveal thickness (CFT) and/or peripapillary edema as measured by spectral domain optical coherence tomography (SD-OCT) in central and/or paracentral fields from Day 0 (Baseline), Day 180 (M6), Day 360 (M12), Day 540 (M18) and 720 (M24)
Mean Change in Choroidal Thickness | Baseline, Month 6, Month 12, Month 18, Month 24
  To determine mean change in choroidal thickness (at fovea) as imaged via EDI-OCT between Day 0 (Baseline), Day 180 (M6), Day 360 (M12), Day 540 (M18), and Day 720 (M24)
Proportion of previously treated and treatment naive patients that require additional dosing outside of the protocol determined dosing schedule | Month 24
  To identify proportion of patients between previously treated and treatment naïve patients that require additional dosing outside of the protocol determined dosing schedule: 3- initial monthly dosing followed by dosing every other month for 720 days (M24)
Assess changes on Autofluorescence | Baseline, Month 6, Month 12, Month 18, Month 24
  To assess changes on autofluorescence (AF) as seen on images from Day 1 (Baseline), Day 180 (M6), Day 360 (M12), Day 540 (M18) and Day 720 (M24)
Incidence and Severity of Ocular and Non-Ocular Adverse Events | Baseline through Month 24
  To determine the incidence and severity of ocular and non-ocular adverse events from Day 1(Baseline) through the end of the study (Day 720)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg T. Kokame, MD, MMS, Principal Investigator — Hawaii Pacific Health
Locations (1):
- Retina Consultants of Hawaii, ‘Aiea, Hawaii, United States

REFERENCES:
- [Derived] Kokame GT, Lai JC, Wee R, Yanagihara R, Shantha JG, Ayabe J, Hirai K. Prospective clinical trial of Intravitreal aflibercept treatment for PolypoIdal choroidal vasculopathy with hemorrhage or exudation (EPIC study): 6 month results. BMC Ophthalmol. 2016 Jul 27;16:127. doi: 10.1186/s12886-016-0305-2. PMID 27465105